CLINICAL TRIAL: NCT00395096
Title: Environmental Exposures, NOS Genes, and Exhaled Nitric Oxide in Pediatric Asthma
Brief Title: Environmental Exposures, Genetics, and Exhaled Nitric Oxide in Pediatric Asthma
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1354; R21HL083145 (NIH); R21HL083145-01A1 (NIH)
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2009-02

CONDITIONS: Asthma
Keywords: Exhaled Nitric Oxide; Asthma; Tobacco Smoke; Allergen
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Asthma is one of the most common childhood diseases. It is chronic and often severely disabling. The amount of nitric oxide that is exhaled while breathing increases with airway inflammation, a symptom of asthma. This study will examine the results from a previous study, the Cincinnati Asthma Prevention (CAP) study, to evaluate the effects of environmental and genetic factors on exhaled nitric oxide (eNO) levels and to determine the relationship between eNO and asthma severity.

DETAILED DESCRIPTION:
Nitric oxide is a naturally occurring gas that plays a role in many body functions. Levels of eNO increase with airway inflammation, a symptom of asthma. Researchers have proposed using eNO as a noninvasive measure to guide physicians in the treatment and medical management of asthma in children. However, more information about eNO is needed before this can happen. This study will perform a secondary analysis of the results from its parent study, the CAP study, which evaluated the effectiveness of preventing asthma in children who had been exposed to environmental tobacco smoke.

This study will not enroll any new participants. Previously collected data from the CAP study will be reevaluated in this study to determine the longitudinal effects of environmental and genetic factors on eNO levels. In addition, the data will be evaluated to determine the relationship between eNO levels and asthma severity. No new data will be collected in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the Cincinnati Asthma Prevention Study
* Diagnosis of asthma
* Lives with someone that smokes at least 5 cigarettes a day

Exclusion Criteria:

* No additional neuromuscular or respiratory disorder that may interfere with safe participation in the parent study
* Does not have electricity
* Plans to move within 1 year of entry into the parent study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cincinnati area children with asthma
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Effects of environmental and genetic factors on exhaled nitric oxide (eNO) levels and the relationship between eNO and asthma severity | Measured through the use of data previously collected in the Cincinnati Asthma Prevention (CAP) study

CONTACTS AND LOCATIONS:
Overall Officials: Adam J. Spanier, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Spanier AJ, Hornung R, Lierl M, Lanphear BP. Environmental exposures and exhaled nitric oxide in children with asthma. J Pediatr. 2006 Aug;149(2):220-6. doi: 10.1016/j.jpeds.2006.04.001. PMID 16887438
- [Result] Wilson SE, Kahn RS, Khoury J, Lanphear BP. Racial differences in exposure to environmental tobacco smoke among children. Environ Health Perspect. 2005 Mar;113(3):362-7. doi: 10.1289/ehp.7379. PMID 15743729